CLINICAL TRIAL: NCT00902733
Title: A Standardized Nursing Intervention Protocol for Pancreatic Cancer as a Chronic Illness
Brief Title: Nurse-Provided Care or Standard Care in Treating Patients With Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marcia Grant, City of Hope Comprehensive Cancer Center
Purpose: Health Services Research
Other Study IDs: 08033; P30CA033572 (NIH); CHNMC-08033; CDR0000629414 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Fatigue; Nausea and Vomiting; Pain; Pancreatic Cancer
Keywords: pain; fatigue; nausea and vomiting; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Fatigue; Nausea; Vomiting; Pain; Pancreatic Neoplasms | interventions — Therapeutics; Psychiatric Rehabilitation

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: fatigue assessment and management
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Meeting with a nurse to assess symptoms and quality of life may be more effective than standard care in treating patients with pancreatic cancer.

PURPOSE: This clinical trial is studying nurse-provided care to see how well it works compared with standard care in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the effects of an advanced practice nurse (APN) standardized nursing-intervention protocol (SNIP) model vs usual care on overall quality of life (QOL) and psychological distress from initial treatment to 6 months post diagnosis for patients with pancreatic cancer.
* To compare symptom control in these patients.
* To compare geriatric assessment outcomes in these patients.
* To test the effects of the SNIP intervention as compared to the usual care group on resource use by these patients.
* To test the effects of SNIP on patients' and clinicians' satisfaction with care.
* To describe the effects of SNIP on patients' management of transitions from one phase of chronic illness to another.
* To identify subgroups of these patients who benefit most from the SNIP in relation to sociodemographic characteristics, disease/treatment factors, and geriatric assessment predictors.
* To obtain feedback from clinicians regarding interpretation of findings and application to the routine care of pancreatic cancer patients.

OUTLINE: Patients are sequentially enrolled to 1 of 2 groups. Group 1 is enrolled during months 4-21 and group 2 during months 25-54.

* Group 1 (usual care): Patient questionnaires are administered at baseline and at 3 and 6 months. The clinicians' satisfaction with care is also evaluated.
* Group 2 (advanced practice nurse [APN] intervention): Patients are accrued by an APN. Patients meet with the APN periodically to assess their physical well-being including ambulatory care needed, care of physical symptoms (i.e., pain, fatigue, nausea and vomiting), and psychological well-being. Questionnaires are administered at baseline and at 3 and 6 months.

In both groups, questionnaires include the FACT-Hep, Memorial Symptom Assessment Scale, Psychological Distress Thermometer, Comprehensive Geriatric Assessment, and Patient Satisfaction with Intervention. Clinicians also complete questionnaires. Patients' medical charts are also reviewed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pancreatic cancer (all stages)

PATIENT CHARACTERISTICS:

* Admitted to City of Hope National Medical Center

  * Resides within a 30-mile radius of the medical center
* No prior cancer

PRIOR CONCURRENT THERAPY:

* No prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Quality of life, psychological distress, symptom relief, geriatric assessment outcome, and resource use at 3 months

SECONDARY OUTCOMES:
Long-term impact at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Grant, RN, DNSc, FAAN, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States